CLINICAL TRIAL: NCT00765895
Title: Nortriptyline for Idiopathic Gastroparesis: A Multicenter, Randomized, Double-Masked, Placebo-Controlled Trial (NORIG)
Brief Title: Nortriptyline for Idiopathic Gastroparesis
Acronym: NORIG
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: U01DK074008 NORIG; 1U01DK073983 (NIH); 1U01DK073975 (NIH); 1U01DK073985 (NIH); 1U01DK074007 (NIH); 1U01DK073974 (NIH); 1U01DK074008 (NIH)
Record Dates: First submitted 2008-10-02; First posted 2008-10-03 (Estimated); Results first posted 2015-04-16 (Estimated); Last update posted 2020-05-14 (Actual); Status verified 2020-04

CONDITIONS: Idiopathic Gastroparesis
Keywords: idiopathic gastroparesis
MeSH Terms: interventions — Nortriptyline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Nortriptyline (Active Comparator): Nortriptyline Hydrochloride dose escalation from 10 mg to 75 mg
  Interventions: Drug: Nortriptyline Hydrochloride
- Placebo (for nortriptyline) (Placebo Comparator): No treatment
  Interventions: Drug: Placebo (for nortriptyline)

INTERVENTIONS:
Drug: Nortriptyline Hydrochloride — Nortriptyline; 10 mg, one capsule, po qhs (by mouth at bedtime each night) x 3 weeks, f03 visit, 25 mg, one capsule, po qhs x 3 weeks, f06 visit, 50 mg, two capsules, po qhs x 3 weeks, f09 visit, 75 mg, three capsules, po qhs x 6 weeks, f15 visit: taper study drug by one capsule a week, off study drug for the last week
  Other Names: Nortriptyline HCl; Pamelor
  Arms: Nortriptyline
Drug: Placebo (for nortriptyline) — Placebo (for nortriptyline), 10 mg, one capsule, po qhs x 3 weeks, f03 visit, 25 mg, one capsule, po qhs x 3 weeks;
  Arms: Placebo (for nortriptyline)

SUMMARY:
The principal objective of this multicenter, randomized, placebo-controlled trial is to evaluate whether treatment with nortriptyline will improve gastroparesis symptoms compared with placebo.

ELIGIBILITY:
Inclusion Criteria:

* Age 21 through 65 years old at registration
* Documentation of delayed gastric emptying on gastric emptying scintigraphy within 2 years of registration, defined as greater than 60% retention at 2 hours or greater than 10% retention at 4 hours
* Symptoms of gastroparesis for at least 6 months (does not have to be contiguous) prior to registration with Gastroparesis Cardinal Symptom Index (GCSI) score of 21 or greater
* Negative upper endoscopy or upper GI series within 2 years of registration

Exclusion Criteria:

* Normal gastric emptying confirmed with scintigraphy
* Diabetic gastroparesis or post-surgical gastroparesis including fundoplication
* Another active disorder which could explain symptoms in the opinion of the investigator
* History of significant cardiac arrhythmias and/or prolonged QTc
* History of seizures
* Use of narcotics more than 3 days per week
* Use of tricyclic antidepressants for refractory symptoms of gastroparesis within 6 weeks prior to randomization
* Use of strongly anticholinergic medications
* Use of calcium channel blockers
* Use of erythromycin
* Clear history of failed trial of nortriptyline use for gastroparetic symptoms
* Symptoms of primary depression or suicidal ideation
* Contraindications to nortriptyline:

  1. hypersensitivity or allergy to any tricyclic antidepressant drug
  2. concomitant therapy with a monoamine oxidase inhibitor (MAOI)
  3. recent myocardial infarction
  4. glaucoma
* Pregnancy or nursing
* Any other condition, which in the opinion of the investigator would impede compliance or hinder completion of the study
* Use of a G tube, J tube,or a central catheter for nutrition
* Use of a gastric electrical stimulator
* Failure to give informed consent

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2009-01 (Actual); Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frank Hamilton, MD, MPH, Study Director — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (7):
- United States (7):
  - California Pacific Medical Center, San Francisco, California
  - Stanford University, Stanford, California
  - University of Michigan Medical Center, Ann Arbor, Michigan
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Texas Tech University Health Sciences Center, El Paso, Texas

IPD SHARING:
Plan to Share IPD: Yes
Data are available at the NIDDK Central Repository: https://repository.niddk.nih.gov/studies/norig/?query=norig
URL: https://repository.niddk.nih.gov/studies/norig/?query=norig

REFERENCES:
- [Derived] Parkman HP, Van Natta ML, Abell TL, McCallum RW, Sarosiek I, Nguyen L, Snape WJ, Koch KL, Hasler WL, Farrugia G, Lee L, Unalp-Arida A, Tonascia J, Hamilton F, Pasricha PJ. Effect of nortriptyline on symptoms of idiopathic gastroparesis: the NORIG randomized clinical trial. JAMA. 2013 Dec 25;310(24):2640-9. doi: 10.1001/jama.2013.282833. PMID 24368464
- See also: Click here for information on gastroparesis research — https://jhuccs1.us/gpcrc/

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: No treatment
  Nortriptyline-Placebo: Nortriptyline-placebo, 10 mg, one capsule, po qhs x 3 weeks, f03 visit, 25 mg, one capsule, po qhs x 3 weeks; f06 visit, 50 mg, two capsules, po qhs x 3 weeks; f09 visit, 75 mg, three capsules, po qhs x 6 weeks, po qhs x 15 wks f15 visit: taper study drug by one capsule a week, off study drug for the last week
Period: Overall Study
Arm/Group | Nortriptyline | Placebo
Started | 65 | 65
Completed | 65 | 65
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nortriptyline | Placebo | Total
Number analyzed (Participants) | 65 | 65 | 130
Age, Continuous [Mean (Standard Deviation); unit: years] | 42 (12) | 40 (12) | 41 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60 | 56 | 116
  Male | 5 | 9 | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 10 | 9 | 19
  White | 54 | 54 | 108
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 8 | 15
  Not Hispanic or Latino | 58 | 57 | 115
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 65 | 65 | 130
Body mass index [Mean (Standard Deviation); unit: kg/m^2] | 27 (5) | 28 (7) | 27 (6)
proton-pump inhibitor taken in last month [Number; unit: participants] — Number of participants reporting that they used a proton-pump inhibitor drug in the last month.
  participants | 48 | 49 | 97
benzodiazepine taken in last month [Number; unit: participants] — Number of participants reporting that they used a benzodiazepine drug in the last month.
  participants | 26 | 14 | 40
prokinetic taken in last month [Number; unit: participants] — Number of participants reporting that they took a prokinetic drug in the last month.
  participants | 23 | 25 | 48
antiemetics taken in last month [Number; unit: participants] — Number of participants reporting that they took an antiemetic drug in the last month.
  participants | 39 | 33 | 72
selective serotonin reuptake inhibitor taken in last month [Number; unit: participants] — Number of participants reporting that they took a selective serotonin receptor reuptake inhibitor drug in the last month.
  participants | 7 | 11 | 18
GSCI total score [Mean (Standard Deviation); unit: units on a scale] — Sum of all 9 GCSI items (sum of nausea, satiety, and bloating subscores). Score ranges from 0-45;higher scores meaning more severe symptoms.
  units on a scale | 30.9 (6.1) | 30.3 (6.5) | 30.6 (6.3)
GSCI- nausea sub score [Mean (Standard Deviation); unit: units on a scale] — Sum of 3 GCSI items: nausea, retching and vomiting symptoms. Each symptom score ranges from 0-5, with a total nausea subscore range from 0-15, with higher scores meaning worse symptom severity.
  units on a scale | 8.2 (3.6) | 8.2 (4.2) | 8.2 (3.9)
GSCI- satiety sub score [Mean (Standard Deviation); unit: units on a scale] — Sum of 4 GSCI items: fullness, not able to finish a normal size meal, feeling excessivley full and loss of appetite symptoms. The sub-score ranges from 0-20, with higher scores meaning worse symptom severity.
  units on a scale | 15.4 (3.4) | 15.1 (4.1) | 15.3 (3.7)
GSCI- bloating sub score [Mean (Standard Deviation); unit: units on a scale] — Sum of 2 GCSI items: bloating and stomach visibly larger symptoms. Each symptom score ranges from 0-5, with a total bloating subscore range from 0-10. Higher scores mean more severe symptoms.
  units on a scale | 7.2 (2.9) | 7.0 (2.7) | 7.1 (2.8)
PAGI-SYM- upper abdominal pain sub score [Mean (Standard Deviation); unit: units on a scale] — Sum of 2 PAGI-SYM items: upper abdominal pain and upper abdominal discomfort symptoms. Each symptom score ranges from 0-5, with a total upper abdominal pain score range from 0-10. Higher scores mean more severe symptoms.
  units on a scale | 6.8 (2.9) | 6.5 (2.9) | 6.6 (2.9)
PAGI-SYM- lower abdominal pain sub score [Mean (Standard Deviation); unit: units on a scale] — Sum 2 PAGI-SYM items: lower abdominal pain and lower abdominal discomfort symptoms. Each symptom score ranges from 0-5, with a total lower abdominal pain score range from 0-10. Higher scores mean more severe symptoms.
  units on a scale | 4.7 (3.3) | 4.3 (3.3) | 4.5 (3.3)
PAGI-SYM- GERD sub score [Mean (Standard Deviation); unit: units on a scale] — Sum of 7 PAGI-SYM items rating heartburn, discomfort in the chest, regurgitation/reflux and bitter acid taste in your mouth symptoms. Each symptom score ranges from 0-5, with a total GERD score range from 0-35. Higher scores mean more severe symptoms.
  units on a scale | 15.4 (9.4) | 17.9 (10.5) | 16.7 (10.7)
GI symptoms constipation sub score [Mean (Standard Deviation); unit: units on a scale] — The constipation symptom score ranges from 0-5, higher scores mean more severe symptoms.
  units on a scale | 2.8 (1.9) | 2.4 (1.7) | 2.6 (1.8)
GI symptom diarrhea sub score [Mean (Standard Deviation); unit: units on a scale] — The diarrhea score ranges from 0-5; higher scores mean more severe symptoms.
  units on a scale | 1.8 (1.7) | 2.0 (1.8) | 1.9 (1.8)
PAGI-SYM nausea/vomiting predominant symptom [Number; unit: participants] — Number of participants reporting either nausea or vomiting as their predominant symptom on the PAGI-SYM.
  participants | 27 | 22 | 49
clinical global patient impression score [Mean (Standard Deviation); unit: units on a scale] — A Clinical Global Patient Impression (CGPI) question quantified overall relief of symptoms. This question asked, "Compared to the way you usually felt before entering the study,how would you rate your relief of symptoms during the past week?" Items coded -3 (very considerably worse) to 3 (completely better). Lower scores mean worsening of symptoms.
  units on a scale | -0.7 (0.9) | -0.7 (1.2) | -0.7 (1.0)
Gastroparesis Symptom Rating Scale score [Mean (Standard Deviation); unit: units on a scale] — Gastrointestinal Symptom Rating Scale (GSRS) assesses gastrointestinal symptoms seen in irritable bowel syndrome and peptic ulcer disease. The mean of 15 items coded 1 (no discomfort) to 7 (very severe discomfort). Higher scores mean worse symptoms.
  units on a scale | 3.6 (1.1) | 3.7 (1.2) | 3.6 (1.2)
SF-36 Quality of Life - Physical component [Mean (Standard Deviation); unit: units on a scale] — he SF-36 consists of scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.
  units on a scale | 35 (10) | 36 (10) | 35 (10)
SF-36 Quality of Life -Mental component [Mean (Standard Deviation); unit: units on a scale] — he SF-36 consists of scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.
  units on a scale | 41 (13) | 40 (13) | 40 (13)
Beck Depression Inventory- total score [Mean (Standard Deviation); unit: units on a scale] — Sum of 21 BDI items coded 0 (absence) to 3 (severe) with a total score range of 0-63. Higher scores mean greater depression symptom severity.
  units on a scale | 17 (11) | 18 (12) | 17 (12)
Beck Depression Inventory- severe depression score [Number; unit: participants] — Number of participants with a total score greater than 28 on the Beck Depression Inventory, or scoring a "2" or "3" on either of two items (pessimism and suicidal thoughts) which are indicative of severe depression.
  participants | 12 | 15 | 27
Brief Pain Inventory- severity score [Mean (Standard Deviation); unit: units on a scale] — Mean of 4 Brief Pain Inventory items, where each item is coded 0 (no pain) to 10 (pain as bad as you can imagine) with higher scores meaning greater pain.
  units on a scale | 4.0 (2.5) | 4.1 (2.7) | 4.0 (2.6)
Brief Pain Inventory- interference score [Mean (Standard Deviation); unit: units on a scale] — Mean of 7 Brief Pain Inventory items where each item is coded 0 (does not interfere) to 10 (completely interferes) with higher scores indicating a higher degree to which pain interferes with daily life.
  units on a scale | 4.2 (3.0) | 4.1 (3.3) | 4.1 (3.1)
State Trait Anxiety Inventory- State Anxiety score [Mean (Standard Deviation); unit: units on a scale] — The STAI measures anxiety - state anxiety, or anxiety about an event. The sum of 20 items coded 1 (not at all) to 4 (very much so) for a total score range of 0-80. Higher scores are positively correlated with higher levels of anxiety.
  units on a scale | 42 (13) | 41 (12) | 42 (12)
State Trait Anxiety Inventory- Trait Anxiety score [Mean (Standard Deviation); unit: units on a scale] — The STAI measures trait anxiety, or anxiety level as a personal characteristic. The sum of 20 items coded 1 (almost never) to 4 (almost always)gives a total score range of 0-80. Higher scores are positively correlated with higher levels of trait anxiety.
  units on a scale | 43 (12) | 43 (13) | 43 (12)
Patient Health Questionnaire-15 [Mean (Standard Deviation); unit: units on a scale] — The Patient Health Questionnaire (PHQ) is a multiple-choice self-report inventory that is used as a screening and diagnostic tool for somatic symptoms. The sum of 15 items coded 0 (not bothered at all) to 2 (bothered a lot); total score range 0-30).Higher scores indicate higher somatic symptoms.
  units on a scale | 14 (5) | 14 (5) | 14 (5)

OUTCOME MEASURES:

1. Primary Outcome: Decrease From the Baseline GCSI of at Least 50% on Any Two Consecutive Follow-up Visits
Description: A decrease from the baseline Gastroparesis Cardinal Symptom Index (GCSI) score (sum of the 9 individual symptom scores) of at least 50% on any two consecutive follow-up visits during the 15 week treatment period with maximum tolerated study drug dose. The total score ranges from 0-45 with higher scores indicating greater symptom severity.
Time Frame: at end of treatment, 15 weeks from baseline assessment
Population: intention to treat
Measure: Number (95% Confidence Interval); unit: participants
Arm/Group | Nortriptyline | Placebo
Number analyzed (Participants) | 65 | 65
participants | 15 [13.5 to 35.2] | 14 [12.3 to 33.5]
Statistical Analysis 1: Comparison: Nortriptyline vs Placebo; Test type: Superiority or Other; p = 0.86, Mantel Haenszel; Stratified by clinic

ADVERSE EVENTS:
Time Frame: Duration of treatment. 15 weeks and for 3 weeks after treatment ended ( 18 weeks total)
Arm/Group | Nortriptyline | Placebo
Serious Adverse Events (participants affected / at risk) | 5/65 | 1/65
Other Adverse Events (participants affected / at risk) | 18/65 | 23/65
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nortriptyline (N=65) | Placebo (N=65)
allergic reaction (General disorders) | 1 (1) | 0 (0)
vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0)
Nausea and vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
cardiac event (Cardiac disorders) | 1 (1) | 0 (0)
abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nortriptyline (N=65) | Placebo (N=65)
Nervous system (Nervous system disorders) | 4 (5) | 2 (2)
gastrointestinal events (Gastrointestinal disorders) | 3 (5) | 5 (6)
cardiac (Cardiac disorders) | 5 (6) | 5 (5)
rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
renal and urinary events (Renal and urinary disorders) | 3 (3) | 0 (0)
ocular events (Eye disorders) | 1 (1) | 0 (0)
swelling of hands and feet (General disorders) | 1 (1) | 0 (0)
psychiatric (Psychiatric disorders) | 0 (0) | 3 (5)
endocrine (Endocrine disorders) | 0 (0) | 1 (1)
weight gain/loss (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
general disorders (General disorders) | 0 (0) | 3 (3) — insomnia
pain (General disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No